CLINICAL TRIAL: NCT03572621
Title: Development and Evaluation of a Therapeutic Education Intervention in Prostate Cancer Patients Treated With Radical Prostatectomy to Improve Their Sexuality
Acronym: PRODUCAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0010
Record Dates: First submitted 2018-06-04; First posted 2018-06-28 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Patients in the experimental group are offered to participate in a 6-session therapeutic education program on sexuality, ranging from 15 days before surgery to approximately 3 months after. This in addition to the current care by the teams of care about sexual rehabilitation (information and medication prescriptions).
  Interventions: Other: Therapeutic education
- Control group (Sham Comparator): Patient without therapeutic education.
  Interventions: Other: Collection of data concerning their sexuality
- Partner (Other): Patient's partner.
  Interventions: Other: Participation

INTERVENTIONS:
Other: Therapeutic education — Patients will benefit from the first session of preoperative therapeutic education, then the next 5 sessions will be done postoperatively over a period of 4 month and a half.
  Session 1: The first session will be devoted appropriately to patient education. It will take place on the day of the preoperative anesthesia consultation.
  Session 2: day of discharge from hospital. Make the patient adhere to the concept of post PR erectile rehabilitation in the same way as sphincter reeducation.
  Session 3: Presentation of available treatments, start intracavernous injections.
  Session 4: Acquisition of know-how on treatment management. Reduce anxiety. Session 5: Encourage the resumption of intercourse very gradually. The presence of the partner will be advised.
  Session 6: measure of the evolution of the representations and knowledge of the patient. The skills of the patient will be evaluated from problem situations, motivation scale. The know-how will be evaluated using observation grid.
  Arms: Experimental group
Other: Collection of data concerning their sexuality — Patients in the control group are offered to participate in the study, which consists of collecting data on their sexuality. This in addition to the current care by the teams of care about erectile rehabilitation (information and medication prescriptions).
  Arms: Control group
Other: Participation — Participation in a therapeutic education day.
  Arms: Partner

SUMMARY:
Prostate cancer is the most common cancer in France (54,000 cases in 2011). About 20,000 radical prostatectomies (PR) per year are performed. Despite the progress of PR over the past 20 years, the rate of erectile dysfunction post PR varies between 30 and 90% and only 16% of operated men recover their pre-treatment erections.

There is currently no validated post-prostatectomy rehabilitation protocol. The associations of patients, including the National Association of Prostate Cancer Patients have a very strong demand for treatment of sexual problems after treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients treated in urology consultation at the University Hospital of Lyon Sud or Edouard Herriot:

* Aged over 18
* presenting a cancerous pathology of the prostate having an indication of radical prostatectomy with or without preservation of the neurovascular strips.
* affiliated to a social security scheme.
* and having been informed and given informed consent to participation in the program.

Exclusion Criteria:

* Refusal of participation, signature of consent,
* protected major patients, under guardianship or curators.
* Patients unable to understand the course of the study
* Patient with a documented history of cognitive or psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients treated in urology consultation at the University Hospital of Lyon Sud or Edouard Herriot Hospital for a Prostatectomy
Enrollment: 240 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change the quality of sexual life of patients treated with radical prostatectomy (PR) | 18 months
  Comparison of the difference in self-Esteem quotation and Relationship (SEAR) questionnaire, between the experimental group and control, between inclusion and Month 18.

SECONDARY OUTCOMES:
Sexual function | Month 1, 6, 12 and 18
  Measure of The International Index of Erectile Function (IIEF-EF) score. This validated score measures the erectile component.
General quality of life | Month 1, 6, 12 and 18
  Signing of questionnaire EuroQol-D5 (EQ-D5)
Sexual quality of life of the partner | Month 1, 6, 12 and 18
  Index of Sexual Life (ISL) questionnaire, validated questionnaire specifically created to assess the impact of erectile dysfunction (ED) in the partner.
Number of erections obtained in the last month | Month 1, 6, 12 and 18
  Patient questionnaire to be filled every month at home by the patient and the partner
Number of reports deemed satisfactory | Month 1, 6, 12 and 18
  Patient questionnaire to be filled every month at home by the patient and the partner
Number of intracavernous injections performed per week | Month18
  Patient questionnaire to be filled every month at home by the patient and the partner
Patient Activation Measure (questionnaire PAM) | Month18
Erection Hardness Score (EHS) | Month 1, 6, 12 and 18
Continence: urinary handicap measurement scale (MHU) | Month 1, 6, 12 and 18
Penis size (cm) | Month 1, 6, 12 and 18
Knowledge acquisition measured by quizz build for the study made of simulated cases | Month 1, 6, 12 and 18
acquisition of sexual intercourse management skills measured by quizz build for the study made of simulated cases | Month 1, 6, 12 and 18
Anxiety level measured by the Hospital Anxiety and Depression (HAD) scale | Month 6 and18
Depression level measured by the Hospital Anxiety and Depression (HAD) scale | Month 6 and18

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Etienne TERRIER, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hôpital Hédouard Herriot, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite